CLINICAL TRIAL: NCT07069101
Title: The Effect of Continuous Erector Spinae Block Versus Continuous Edge of Laminar Block on The Quality of Analgesia and Diaphragmatic Excursion in Patients With Multiple Rib Fractures. A Prospective Randomized Trail.
Brief Title: Continuous Erector Spinae Block Versus Continuous Edge of Laminar Block on The Quality of Analgesia and Diaphragmatic Excursion in Patients With Multiple Rib Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Abdel Hamid Muhammed, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine Department, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD297/10/24
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Erector Spinae Block; Edge of Laminar Block; Analgesia; Diaphragmatic Excursion; Multiple Rib Fractures
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae group (Experimental): Patients will receive continuous ipsilateral erector spinae plane block.
  Interventions: Other: Erector spinae block
- Edge of lamina group (Experimental): Patients will receive continuous ipsilateral edge of laminar block.
  Interventions: Other: Edge of lamina block

INTERVENTIONS:
Other: Erector spinae block — Patients will receive continuous ipsilateral erector spinae plane block.
  Arms: Erector spinae group
Other: Edge of lamina block — Patients will receive continuous ipsilateral edge of laminar block.
  Arms: Edge of lamina group

SUMMARY:
This prospective randomized clinical trial aims to compare the effect of continuous erector spinae plane block versus continuous edge of laminar block on the quality of analgesia and diaphragmatic excursion in patients with unilateral traumatic multiple rib fractures.

DETAILED DESCRIPTION:
Rib fractures occur in up to 12% of all trauma patients, most commonly due to blunt thoracic trauma, and pose a significant health care burden with their associated morbidity and mortality.

The erector spinae plane block (ESB) is a myofascial plane technique in which a needle is inserted under ultrasound guidance deep to the erector spinae muscle group, allowing an infusion of local anesthetic to diffuse to both the dorsal and ventral rami of the spinal nerves, thereby supplying the rib cage. This technique can be used as a single-shot method or to facilitate the placement of a catheter, allowing for continuous infusion and/or intermittent bolus to provide long-lasting analgesia.

The edge of laminar block (ELB) is a novel technique in which local anesthetics are injected at the lateral edge of the lamina. It has been proven to provide sensory analgesia during rib fractures.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21 and 65 years.
* Both sexes.
* With unilateral traumatic multiple fracture ribs (≥ 3), admitted to the surgical intensive care unit within the first day of trauma.

Exclusion Criteria:

* Patients' rejection.
* Body mass index ≥ 35 (kg/m2).
* Bleeding and Coagulation disorders.
* Known hypersensitivity to the study drugs.
* Vertebral deformity.
* Respiratory, cardiac, renal or hepatic dysfunction.
* Patients with major trauma involving extra-thoracic structures (e.g., head, spine, pelvis, and abdominal visceral injuries).
* Mental or cognitive dysfunction,
* History of chronic analgesic or drug abuse.
* Local infection at the site of the block.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 4 days postoperatively
  If the Numeric Rating Scale (NRS) is 4 or more IV morphine 3mg will be given.

SECONDARY OUTCOMES:
Degree of pain | 4 days postoperatively
  The degree of pain will be assessed using the Numeric Rating Scale (NRS) at rest and on coughing will be assessed before the block, at 60 minutes after the block, and then every 8 hours for 4 days.
Diaphragmatic excursion | 4 days postoperatively
  Diaphragmatic excursion will be assessed before the block, at 60 minutes after the block, and then every 8 hours for 4 days.
Incidence of adverse events | 4 days postoperatively
  Incidence of adverse events such as hematoma, local anesthetic systemic toxicity, respiratory complications, pneumothorax, nausea, and vomiting.
Forced vital capacity | 4 days postoperatively
  Forced vital capacity (FVC) will be assessed before the block, at 60 minutes after block, and then every 8 hours for 4 days.
Forced expiratory volume 1 | 4 days postoperatively
  Forced expiratory volume 1 (FEV1) will be assessed before the block, at 60 minutes after block, and then every 8 hours for 4 days.
Forced expiratory volume 1 (FEV1)/Forced vital capacity (FVC) | 4 days postoperatively
  Forced expiratory volume 1 (FEV1)/Forced vital capacity (FVC) will be assessed before the block, at 60 minutes after block, and then every 8 hours for 4 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.